CLINICAL TRIAL: NCT04799626
Title: Population Pharmacokinetics and Dosage Individualization of Biapenem,Meropenem,Piperacillin and Tazobactam,Tigecycline,Levofloxacin .Etc in Elderly Patients Who Was Hospitalized in Intensive Care Unit
Brief Title: Population Pharmacokinetics and Dosage Individualization of Antibiotics in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: The Second Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacoligy, Shandong University
Other Study IDs: 2021-Antibiotics-009
Record Dates: First submitted 2021-03-14; First posted 2021-03-16 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Elderly Infection
Keywords: biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin.etc; elderly ICU patients; dosage regimen; pharmacokinetics and pharmacodynamics
MeSH Terms: interventions — biapenem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment: The use of antimicrobial agents depends on the clinical practice.
  Interventions: Drug: biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin.etc

INTERVENTIONS:
Drug: biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin.etc — biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin.etc extended infusion time or continuous infusion for 24 hours;Tigecycline changed standard does for treatment.

SUMMARY:
The investigator's purpose is to study the pharmacokinetics and pharmacodynamics of biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin.etc in elderly ICU patients and recommend an individual dosage regimen of those antibiotics.

DETAILED DESCRIPTION:
The use of biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin.etc in elderly ICU patients during clinical treatment depended mostly on experience. Besides, there was no recommended dose for elderly patients in drug instruction, Therefore, we aim to study the pharmacokinetics and pharmacodynamics in elderly ICU patients and provide a tailormade regimen.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥65 years old; (2) According to the doctor's advice, use biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin.etc for anti-infection treatment;

Exclusion Criteria:

* (1) Patients who are expected to die within 48 hours; (2) Patients with allergic to β-lactam antibiotics, Carbapenems, Ticacycline and Levofloxacin.etc drugs; (3) Patients receiving other investigational drugs; (4) Other factors that the researcher considers unsuitable for inclusion.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly ICU patients (≥65years）treated with biapenem,meropenem,piperacillin and tazobactam,tigecycline and levofloxacin.etc who was hospitalized in the Second Hospital of Shandong University.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The peak plasma drug concentration of biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin.etc | at (5-10) minutes after intravenous administration
  To detect the peak plasma drug concentration of biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin.etc after intravenous administration.
The random plasma drug concentration of biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin.etc | at (0.5-10) hours after intravenous administration
  To detect the random plasma and cerebrospinal fluid drug concentration of biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin after intravenous administration.
The trough plasma drug concentration of biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin.etc | at 1-2 hours before the next administration
  To detect the trough plasma drug concentration of biapenem,meropenem,piperacillin and tazobactam,tigecycline,levofloxacin after intravenous administration.

SECONDARY OUTCOMES:
C-reaction protein | Through study completion, an average of 14 days
  Blood routine examination
level of procalcitonin | Through study completion, an average of 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Ph.D, Study Chair — The Second Hospital of Shandong University
Locations (1):
- Wei Zhao, Jinan, Shandong, China